CLINICAL TRIAL: NCT01016574
Title: Evaluating the Adequacy of Giro-Couch to Support Prone Breast Boost Irradiation Using Intensity Modulated Radiation Therapy(IMRT)Technique With Image-guided Radiation Therapy(IGRT).
Brief Title: Evaluating the Adequacy of Giro-Couch to Support Prone Breast Boost Irradiation Using IMRT Technique With IGRT.
Acronym: IN902
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azimuth Therapy Ltd. (Industry)
Responsible Party: Merav Ben-David, M. D., Institute of Oncology , The Chaim Sheba Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7326-09-SMC
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- women with stage I or II breast cancer (Other)
  Interventions: Device: Support Device for Prone radiation therapy (Giro-Couch)

INTERVENTIONS:
Device: Support Device for Prone radiation therapy (Giro-Couch) — Boost irradiation is applied to the ipsilateral breast in eight fractions of 2Gy/Fx

SUMMARY:
The purpose of this study is to evaluate the Giro-couch, an innovative patient support device for the application of prone RT for treatment of breast cancer. This study will assess the feasibility of a new positioning approach to facilitate the delivery of external beam, delivered to the lumpectomy cavity, (the boost dose, partial breast therapy).

DETAILED DESCRIPTION:
Treatments are applied with the subject in the supine position, in ~50 Gy per treatment (~2GY per fraction), over a period of five to six weeks. Energy in use is usually 6-15MV photons. Following the whole breast irradiation, a boost dose is given to the lumpectomy cavity, in order to further reduce the local recurrences in the immediate vicinity of the treated breast. The boost dose is usually applied with electrons, 6-18MEV. Sixteen Gy is the usual dose, 2 Gy/Fx, for 8 fractions.

ELIGIBILITY:
Inclusion Criteria:

Women who satisfy all of the following conditions are the only patients who will be eligible for this study:

* The patient must consent to be in the study and must have signed an approved consent form conforming to federal and institutional guidelines.
* Patients must be ≥ 40 years old.
* The patient must have stage I or II breast cancer. If stage II, the tumor size must be 3 cm or less.
* Surgical treatment of the breast must have been lumpectomy. The margins of the resected specimen must be at least 2mm. Re-excision of surgical margins is permitted.
* Gross disease must be unifocal.
* The target lumpectomy cavity must be clearly delineated and the target lumpectomy cavity/whole breast reference volume must be ≤ 30% based on the treatment planning CT scan.
* The lumpectomy cavity must be delineated with surgical clips by the surgeon.
* Patients are eligible if, based on the postoperative/ simulation CT scan, prone boost RT is judged to be technically deliverable by a prone breast IMRT-IGRT technique.
* Patients with a history of non-breast malignancies are eligible if they have been disease-free for 5 or more years prior to randomization and are deemed by their physician to be at low risk for recurrence. Patients with the following cancers are eligible if diagnosed and treated within the past 5 years: carcinoma in situ of the cervix, carcinoma in situ of the colon, melanoma in situ, and basal cell and squamous cell carcinoma of the skin.

Exclusion Criteria:

* Men are not eligible for this study. Women with one or more of the following conditions also are ineligible for this study.
* T0, T2 (> 3.0 cm), T3, stage III, or stage IV breast cancer (see Appendix A for TNM nomenclature and staging).
* Suspicious microcalcifications, densities, or palpable abnormalities (in the ipsilateral or contralateral breast) unless biopsied and found to be benign.
* Non-epithelial breast malignancies such as sarcoma or lymphoma.
* Proven multicentric carcinoma (invasive cancer or DCIS) in more than one quadrant or separated by 4 or more centimeters.
* Paget's disease of the nipple.
* Synchronous bilateral invasive or non-invasive breast cancer.
* Surgical margins that cannot be microscopically assessed or are positive at pathologic evaluation. (If surgical margins are rendered free of disease by re-excision, the patient is eligible.)
* Clear delineation of the extent of the target lumpectomy cavity not possible.
* Breast implants.
* Prior breast or thoracic RT for any condition
* Collagen vascular disease, specifically dermatomyositis, systemic lupus erythematosis, or scleroderma.
* Pregnancy or lactation at the time of proposed randomization. Women of reproductive potential must agree to use an effective non-hormonal method of contraception during therapy.
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Ease of use and Comfort scale 1-5 | Treatment Day 1 and Treatment Day 8
  The endpoints will be assessed at the conclusion of the subject's first treatment on Treatment Day 1, and at the conclusion of the subject's treatment on Treatment Day 8. Thus the time frame for the Primary Outcome Measure for each subject is 1-8 days.

SECONDARY OUTCOMES:
Dosimetric evaluation | Treatment Day 1, Treatment Day 2, Treatment Day 3, Treatment Day 4, Treatment Day 5, Treatment Day 6, Treatment Day 7, Treatment Day 8
  A Dosimetric evaluation will be performed for each subject, each and every day of subjects's treatment.
Localization time | Treatment Day 1, Treatment Day 2, Treatment Day 3, Treatment Day 4, Treatment Day 5, Treatment Day 6, Treatment Day 7, Treatment Day 8
  The time required for target localization will be performed each and every day of each subject's treatment.
Treatment time | Treatment Day 1, Treatment Day 2, Treatment Day 3, Treatment Day 4, Treatment Day 5, Treatment Day 6, Treatment Day 7, Treatment Day 8
  The time required to apply the prescribed treatment (beam on to beam off).

CONTACTS AND LOCATIONS:
Locations (1):
- The Chaim Sheba Medical Center, Tel Litwinsky, Israel